CLINICAL TRIAL: NCT01356433
Title: Effect of Oral Vitamin C on The Inflammatory Biomarkers in Hemodialysis
Brief Title: Influence of Oral Vitamin C Supplement on the Inflammation Status in Dialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Li Zuo, Renal Division, Department of Medicine, Peking University First Hospital, Peking University First Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: d2a3scvr
Record Dates: First submitted 2011-05-16; First posted 2011-05-19 (Estimated); Last update posted 2012-09-21 (Estimated); Status verified 2012-09

CONDITIONS: Uremia; Inflammation
Keywords: dialysis,inflammation,vitamin C
MeSH Terms: conditions — Uremia; Inflammation | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- arm1, vitamin C treated first (Other): Arm 1(50cases): intervention with oral vitamin C 200mg per day in the first 3 months, then stop oral VitC for the next 3 months.
  Interventions: Drug: oral vitamin C
- Arm 2 control first (Other)
  Interventions: Drug: oral vitamin C

INTERVENTIONS:
Drug: oral vitamin C — cross-over study,2 arms Arm 1(50cases): is given oral vitamin C 200mg per day in the first 3 months, then stop oral VitC for the next 3 months.
  Arm 2(50cases): is not given vitamin C in the first 3 months, then switch to receive oral VitC 200mg per day in the next 3 months.
  Other Names: ascorbic acid
Drug: oral vitamin C — Arm 2(50cases): is not given vitamin C in the first 3 months, then switch to receive oral VitC 200mg per day in the next 3 months.
  Other Names: ascorbic acid

SUMMARY:
Subclinical inflammation is a common phenomenon in patients receiving maintenance hemodialysis (MHD). This is because various pro-inflammatory cytokines are promoted due to metabolic acidosis, volume overload, and / or non-sterile dialysate.

As important antioxidants, vitamin C was prominently consumed by oxidative stress and inflammation. So patients receiving dialysis therapy usually had a low plasma vitamin C level.

It was documented that inflammation was associated with increased risk of cardiovascular morbidity and mortality in patients on dialysis. But the relationship between plasma Vitamin C and each of inflammatory markers and prealbumin was lacking. Because vitamin C had anti-inflammation effect on behalf of its electron receiving ability, the investigators made a hypothesis that vitamin C supplementation can reduce inflammation status in patients on maintenance dialysis

DETAILED DESCRIPTION:
Objective A cross-over study is designed to elucidate if oral vitamin C supplementation can reduce inflammation status in maintenance dialysis patients with low vitamin C level and high CRP level.

Patients, Methods and Expected results Patients About 100 dialysis patients were recruited. Patients will be divided into two groups, and will be followed for at least 6 months.

Methods Arm 1(50cases): is given oral vitamin C 200mg per day in the first 3 months, then stop oral VitC for the next 3 months.

Arm 2(50cases): is not given vitamin C in the first 3 months, then switch to receive oral VitC 200mg per day in the next 3 months.

The demographics were recorded. Plasma Vitamin C was measured by high-performance liquid chromatography. Serum albumin, prealbumin, high-sensitivity C-reactive protein (hsCRP), ferritin, hemoglobin will be measured.

Expected results There may be positive effect of vitamin C supplementation on inflammation in maintenance dialysis patients with vitamin C deficiency and high CRP level.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving maintenance hemodialysis or continuous ambulatory peritoneal dialysis, and dialysis vintage more than 3 months
* Patients aged between 18 and 80 years older
* VitC < 4ug/ml and hsCRP > 3mg/L
* for HD patients, Kt/V > 1.2 per session, at least 3 sessions per week, 4 hours per session
* for PD patients, Kt/V > 1.7 per week
* age and gender matched health control

Exclusion Criteria:

* Active autoimmune disease, malignancy, hepatitis
* Positive HIV serology
* Any kind of acute infection within one month, chronic infection
* Currently using steroids or immune-suppressants
* Pregnancy or breast feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
the level of hsCRP | 6 months

SECONDARY OUTCOMES:
the level of prealbumin | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Li Zuo, MD, Study Director — Renal Division, Department of Medicine, Peking University First Hospital, Beijing, China
Locations (1):
- hemodialysis center of Renal Division, Department of Medicine, Peking University First Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Colombijn JM, Hooft L, Jun M, Webster AC, Bots ML, Verhaar MC, Vernooij RW. Antioxidants for adults with chronic kidney disease. Cochrane Database Syst Rev. 2023 Nov 2;11(11):CD008176. doi: 10.1002/14651858.CD008176.pub3. PMID 37916745
- [Derived] Zhang K, Li Y, Cheng X, Liu L, Bai W, Guo W, Wu L, Zuo L. Cross-over study of influence of oral vitamin C supplementation on inflammatory status in maintenance hemodialysis patients. BMC Nephrol. 2013 Nov 14;14:252. doi: 10.1186/1471-2369-14-252. PMID 24228847